CLINICAL TRIAL: NCT07378098
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Parallel, Phase 3 Study to Evaluate the Efficacy and Safety of KLH-2109 in Patients With Uterine Fibroids and Menorrhagia
Brief Title: to Evaluate the Efficacy and Safety of KLH-2109 in Patients With Uterine Fibroids and Menorrhagia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JW25301
Record Dates: First submitted 2026-01-19; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Menorrhagia; Uterine Fibroids
Keywords: Uterine Fibroids; Menorrhagia
MeSH Terms: conditions — Menorrhagia; Leiomyoma

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, active-controlled, parallel, phase III
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KLH-2109+ Leurprorelin acetate Placebo (Experimental): KLH-2109: 200mg/day for 24 weeks(PO, QD) Leurprorelin acetate Placebo: Once every 4 weeks, subcutaneous injection
  Interventions: Drug: KLH-2109+ Leurprorelin acetate Placebo
- KLH-2109 Placebo + Leurprorelin acetate (Active Comparator): KLH-2109 Placebo: 24 weeks(PO, QD) Leurprorelin acetate : 1.88mg or 3.75mg, Once every 4 weeks, subcutaneous injection
  Interventions: Drug: KLH-2109 Placebo + Leurprorelin acetate

INTERVENTIONS:
Drug: KLH-2109+ Leurprorelin acetate Placebo — KLH-2109 200mg/day for 24 weeks(PO, QD) Leurprorelin acetate Placebo: Once every 4 weeks, subcutaneous injection
  Other Names: KLH-2019+ Leurprorelin acetate Placebo
  Arms: KLH-2109+ Leurprorelin acetate Placebo
Drug: KLH-2109 Placebo + Leurprorelin acetate — KLH-2109 Placebo: for 24 weeks(PO, QD) Leurprorelin acetate Placebo: 1.88mg or 3.75mg , Once every 4 weeks, subcutaneous injection
  Other Names: KLH-2019 Placebo + Leurprorelin acetate Placebo
  Arms: KLH-2109 Placebo + Leurprorelin acetate

SUMMARY:
The goal of this clinical trial was to determine whether the investigational drug KLH-2109 is effective for treating excessive menstrual bleeding in patients with uterine fibroids. Uterine fibroids are benign tumors that grown in the uterus.

The primary objectives of this trial were to answer the following questions:

* Does KLH-2109 lower the amount of menstrual bleeding?
* Does KLH-2109 reduce menstrual bleeding?
* Is KLH-2109 safe for participants to use?

Investigators will compare KLH-2109 with a standard of care treatment (control) to determine which treatment is more effective.

Participants will be required to follow:

* Take either KLH-2109 or the common treatment as a pill
* Visit the clinic regularly for health checkups and safety tests
* Keep track of their bleeding and any health changes during the study

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-blind, Active-controlled, Parallel, Phase 3

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with uterine fibroids

Exclusion Criteria:

* Metrorrhagia or anovulatory bleeding
* Patients with a history of total hysterectomy or bilateral oophorectomy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Uterine fibroid patients with menorrhagia
Enrollment: 254 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a total PBAC score < 10 | Week 6 to the day before Week 12
  Proportion of subjects with a total PBAC score < 10 from Week 6 to the day before Week 12 after administration of the investigational product

SECONDARY OUTCOMES:
Proportion of subjects with a total PBAC score < 10 | Week 6 , Week12, Week 18, Week 24
  Proportion of subjects with a total PBAC score < 10 from Week 2 to the day before Week 6 after administration of the investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Yeol Park, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No